CLINICAL TRIAL: NCT02409524
Title: Phase IIA Clinical Study Of An Individualized Anti-Cancer Vaccine (CRCL-ALLOVAX) in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: An Individualized Anti-Cancer Vaccine in Advanced Hepatocellular Carcinoma Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-022-HCC-BKK-VAX+S
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2017-11

CONDITIONS: Advanced Adult Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): The treatment schedule of AlloVax includes: (1) Priming segment with ID injections of AlloStim on Days 0, 3, 7 and 10. (2) Vaccination segment with ID injections of AlloStim+CRCL on Days 14, 17, 21 and 24. (3) Activation segment with IV push infusion of AlloStim on Day 28. (4) Booster Segment with monthly (every 28 days) ID injections of CRCL alone beginning on Day 56. These injections will continue until all the vaccine is used or the death of the subject
  Interventions: Biological: AlloVax; Biological: AlloStim; Biological: CRCL

INTERVENTIONS:
Biological: AlloVax — Personalized anti-cancer vaccine (injection of AlloStim followed immediately by the injection of CRCL)
  Other Names: CRCL and AlloStim
Biological: AlloStim — AlloStim (ID) injection AlloStim (IV) infusion
  Other Names: AlloStim ID; AlloStim IV
Biological: CRCL — Autologous tumor-derived chaperone protein mixture
  Other Names: Chaperone Rich Cell Lysate

SUMMARY:
This is an open-label, single site, Phase IIA clinical trial to investigate the safety and efficacy of an individualized anti-cancer vaccine (CRCL-AlloVax) in advanced HCC patients.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) or primary liver cancer is the third leading cause of cancer death worldwide. It accounts for 90% of all liver cancers. More than 80% of patients present with advanced or unresectable disease.

For patients with vascular invasion and/or metastases, the only approved therapy that offers a survival advantage is Sorafenib (Nexavar®). While palliative systemic chemotherapy other than Sorafenib is sometimes offered for HCC, there is no evidence that any chemotherapy has any meaningful therapeutic benefit, especially in overall survival. Subjects in the current study will either have completed at least 90 days of sorafenib treatment or are not able to receive sorafenib due to intolerability or unable to afford. Subjects will continue sorafenib as tolerated while receiving experimental therapy. The experimental dosing schedule has four segments: (1) priming, which consists of intradermal AlloStim alone; (2) vaccination, which consists of intradermal dosing of AlloStim+CRCL; (3) activation, which consists of an intravenous infusion of AlloStim; and (4) booster, which consists of monthly intradermal injections of CRCL alone

ELIGIBILITY:
Inclusion criteria:

1. Males and females who are at least 18 years of age at time of enrollment
2. Histologically confirmed hepatocellular carcinoma with or without positive HBV and/or HCV, not candidate for local regional intervention
3. Minimum of 90 days of sorafenib treatment or ineligible for sorafenib
4. Child-Pugh Stage A-B (score ≥ 5 and ≤ 9)
5. Performance status: ECOG < 2 with no deterioration over the previous 2 weeks
6. Measurable disease (for mRECIST)
7. Lesion amenable for percutaneous tumor harvest and follow up biopsy
8. Adequate bone marrow, liver and renal function as assessed by the following:

   * Hemoglobin > 10.0 g/dl
   * Absolute neutrophil count (ANC) > 1,500/mm3
   * Platelet count > 75,000/μl
   * ALT and AST < 2.5 x ULN
   * Alkaline phosphatase < 4 x ULN
   * Serum creatinine < 1.5
9. Women of child-bearing potential: negative pregnancy test
10. Patients of child producing potential: usage of contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental product
11. Ability to understand the study, its inherent risks, side effects and potential benefits and ability to give written informed consent to participate

Exclusion criteria:

1. Severe ascites, massive or uncontrolled (+3 on Child-Pugh calculator)
2. Severe encephalopathy, uncontrolled (+3 on Child-Pugh calculator)
3. INR > 1.5
4. Participation in another clinical trial evaluating experimental treatments or procedures or receiving medication/treatment for HCC other than sorafenib
5. Any autoimmune disorder
6. Any clinical condition requiring systemic steroids or current immunosuppressive therapy, including: cyclosporine, antithymocyte globulin, or tacrolimus within 1 month of study entry
7. HIV positive or syphilis
8. History of cardiac disease: congestive heart failure > NYHA class 2; cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or Digoxin are permitted) or uncontrolled hypertension
9. Active clinically serious infections (> grade 2 NCI-CTCAE version 4.0)
10. History of organ or tissue allograft
11. Advanced liver cirrhosis
12. Interferon or thalidomide within 1 month prior to signing informed consent
13. Uncontrolled concurrent serious medical or psychiatric illness
14. Clinically apparent central nervous system metastases or carcinomatous meningitis
15. History of blood transfusion reactions
16. Known allergy to murine monoclonal antibodies or bovine products or cow milk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
To evaluate survival compared to historical controls | Approximately 12 months
  Baseline to date of death from any cause

SECONDARY OUTCOMES:
To assess AFP as surrogate end-point for response and/or survival | Approximately 6 months
  Biomarker concentration will be evaluated at different time points
To assess mRECIST as surrogate end-point for response and/or survival | Approximately 6 months
  Objective tumor responses by mRECIST will be compared with OS
To evaluate safety in advanced HCC (adverse events) | Approximately 6 months
  Subjects will be followed by physical exam, blood labs, CT scan and biopsy for any adverse events

OTHER OUTCOMES:
Anti-Tumor Response | 30 days
  Correlation of radiographic tumor burden assessment (mRECIST) with actual tumor burden determined by histological examination of biopsy samples
Tumor-Specific Immunity | 30 days
  Immunological end-points as surrogate markers of response and/or survival

CONTACTS AND LOCATIONS:
Overall Officials: Wirote Lausoontornsiri, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute of Thailand Address: 268/1 Rama Rd. Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No